CLINICAL TRIAL: NCT04077801
Title: Biomechanical Changes in Women With Post-partum Pelvic Girdle Pain: An Observational Case-control Study
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, rovan mohamed saad elbesh, doctor, Misr University for Science and Technology
Other Study IDs: P.T.REC/012/005284
Record Dates: First submitted 2019-09-01; First posted 2019-09-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Postpartum Pain
Keywords: Pelvic girdle Pain, lumbopelvic angles, pelvic parameters, and temporomandibular joint disorders.
MeSH Terms: conditions — Pelvic Girdle Pain; Temporomandibular Joint Disorders | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group (group A): Maximal vertical mouth opening (MIO):
  From sitting position, with the use of the calliper, the distance between the incisal edges along the midline of the upper and lower central incisors without pain was measured, by placing one end of the poley gauge against the incisal edge of one of the upper central incisors, and the other end against the incisal edge of the opposing lower incisor.
  The distance recorded in millimetres, the subjects was instructed to" open your mouth as wide as possible without causing pain or discomfort". The poley gauge was sterilized with antiseptic solution before and after each measure Postpartum pain Intervention 'Visual analogue scale'
  Interventions: Diagnostic Test: diagnostic test; Diagnostic Test: Postpartum pain; Other: Visual analogue scale
- Control group (group B):: Maximal vertical mouth opening (MIO):
  From sitting position, with the use of the calliper, the distance between the incisal edges along the midline of the upper and lower central incisors without pain was measured, by placing one end of the poley gauge against the incisal edge of one of the upper central incisors, and the other end against the incisal edge of the opposing lower incisor.
  The distance recorded in millimetres, the subjects was instructed to" open your mouth as wide as possible without causing pain or discomfort". The poley gauge was sterilized with antiseptic solution before and after each measure Postpartum pain Intervention 'Visual analogue scale'
  Interventions: Diagnostic Test: diagnostic test; Diagnostic Test: Postpartum pain; Other: Visual analogue scale

INTERVENTIONS:
Diagnostic Test: diagnostic test — diagnostic test
Diagnostic Test: Postpartum pain — test
Other: Visual analogue scale — test TMJ /pelvic angle/lumber angle

SUMMARY:
Research suggests that changes in pelvic alignment during the perinatal period are the primary cause of pelvic girdle pain (PGP), both perinatally and postnatally. Researchers also report an association between temporomandibular joint disorder (TMD) and changes in lumbopelvic alignment. There are, however, no reports investigating temporomandibular joint disorders or changes in biomechanical alignment among women with postpartum pelvic girdle pain.

DETAILED DESCRIPTION:
Research suggests that changes in pelvic alignment during the perinatal period are the primary cause of pelvic girdle pain (PGP), both perinatally and postnatally. Researchers also report an association between temporomandibular joint disorder (TMD) and changes in lumbopelvic alignment. There are, however, no reports investigating temporomandibular joint disorders or changes in biomechanical alignment among women with postpartum pelvic girdle pain.

ELIGIBILITY:
Inclusion Criteria:

- The age of the participants will be ranged from 20 to 40 years. Their body mass index will be ranged from 20 to 25 kg/m2. They will have regular menstrual cycle. They will not receive any hormonal therapy or taking any regular drugs

Exclusion Criteria:

* Bone disease. Discogenic state with radiculopathy or not. Systemic disease of musculoskeletal system. Any sensory problems. Previous vertebral fractures. Major spinal structural abnormality. Major jaw abnormality. Any jaw orthotics or prosthesis. Missing teeth.

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: 75 women will participate in this study, The selected cases divide into a study group(A) included 44 women who have CPP and group (B) included 31 women of the participants were normal and considered the control group. They will be selected from outpatient clinic of obstetrics and Gynaecology department in El-Hosary family health Centre.
  All participants will be given a full explanation of the protocol of the study and informed consent form will be signed from each subject before participating in the study (
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-09-08 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
body mass index | 3 months
  BMI in kg/m^2
Pelvic tilt in degrees: | 3 months
  The blocks are released and the rods are placed over the crest of the ilium. The blocks are then pressed firmly toward the midline. Read the angle from the level. If the gauge reads over 21/2°, the result is listed as positive.Anterior pelvic tilting angle: PALM was used for measuring pelvic tilting angle. A mark was put on a point just inferior to ASIS; another mark was put just inferior to PSIS. The callipers of the PALM were put on these two points
jaw movement | 3 months
  lateral deviation mouth opening (MIO):
  From sitting position, with the use of the calliper, the distance between the incisal edges along the midline of the upper and lower central incisors without pain was measured, by placing one end of the poley gauge against the incisal edge of one of the upper central incisors, and the other end against the incisal edge of the opposing lower incisor.
  The distance recorded in millimeters, the subjects was instructed to" open your mouth as wide as possible without causing pain or discomfort". The poley gauge was sterilized with antiseptic solution before and after each measure
Spinal curves Measurement | 3 months
  lumber angle-pelvic inclination by mm
Satisfaction assessed by the VAS | 3 months
  Degrees of pain will be assessed using a VAS, which was a method of representing subjects' pain on a 10 cm linear scale. Score of 0 meant 'no pain' and 10 meant 'worst pain'. Tomeasure specific symptoms, such as the s

CONTACTS AND LOCATIONS:
Locations (1):
- Rovan Elbesh, Giza, Egypt